CLINICAL TRIAL: NCT03696641
Title: Clinical Assessment of Color Stability and Patient Satisfaction for Polished Versus Glazed Lithium Disilicate Glass Ceramic Restorations and Patient Satisfaction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rasha Sayed Mosallam, Assistant lecturer- fixed prosthodontics department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-09-25
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Color Change of Lithium Disilicate Crowns

STUDY DESIGN:
Who Masked: Participant
Masking Description: participant, outcome assessor double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- glazed IPS e.max (Active Comparator): lithium disilicate glazed crowns that proved to have a good color stability
  Interventions: Other: glazed lithium disilicate crowns; Other: polished lithium disilicate crowns
- polished IPS e.max (Experimental): polished lithium disilicate crowns with the polishing kit
  Interventions: Other: glazed lithium disilicate crowns; Other: polished lithium disilicate crowns

INTERVENTIONS:
Other: glazed lithium disilicate crowns — glazing of IPS e.max crowns
  Other Names: glazed IPS e.max
Other: polished lithium disilicate crowns — polishing of IPS e.max crowns
  Other Names: polished IPS e.max

SUMMARY:
Dental overglaze is consist of colorless glass powder and applied to the fired crown surface to provide a glossy surface,Adjustment procedure break the production of the glaze layer through a natural glaze or overglaze process and create a rough surface, glazing or polishing after adjustment procedures is important to enhance the appearance of the restoration

DETAILED DESCRIPTION:
Dental overglaze is consist of colorless glass powder and applied to the fired crown surface to provide a glossy surface. Natural glaze is a vitrified layer that is formed on the surface of the porcelain containing a glass phase when the porcelain is heated to a glazing temperature for a specific time, Adjustment procedure break the production of the glaze layer through a natural glaze or overglaze process and create a rough surface, The color of porcelain restorations is affected by surface roughness because rough surface reflects light irregularly and less than a glazed surface . Therefore, glazing or polishing after adjustment procedures is important to enhance the appearance of the restoration .

Although glazed surfaces appeared whiter, the CIE L* value measured with the specular component excluded (SCE) geometry was lower than that of polished surfaces (28).Several reports have investigated different polishing techniques that support the use of polishing as an alternative for glazing of ceramic restorations .

Polishing can reduce chair time, eliminates laboratory procedures, infection control may be obtained . Polishing is also important for the porcelain surface for esthetic so several different techniques have been described for repolishing porcelain surfaces in the mouth .

ELIGIBILITY:
Inclusion Criteria:

* All subjects are required to be:

  1. From 18-50 years old, be able to read and sign the informed consent document.
  2. Physically and psychologically able to tolerate conventional restorative procedures
  3. have no active periodontal or pulpal diseases, have teeth with good restorations
  4. Willing to return for follow-up examinations and evaluation

Exclusion Criteria:

* 1. Patients in the growth stage with partially erupted teeth 2. Patients with poor oral hygiene and motivation 3. Pregnant women's 4. Psychiatric problems or unrealistic expectations

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
color stability | one year
  L* a* b* values and ∆E

SECONDARY OUTCOMES:
patient satisfaction | one year
  patient satisfaction through a questionnaire

IPD SHARING:
Plan to Share IPD: No